CLINICAL TRIAL: NCT05118048
Title: CLIA Waived Study: StatStrip Lactate, Hemoglobin, and Hematocrit Meter in Whole Blood
Brief Title: StatStrip Lactate, Hemoglobin, and Hematocrit Meter in Whole Blood
Status: Terminated | Type: Observational
Why Stopped: Patient recruitment too slowly
Sponsor: Nova Biomedical (Industry)
Collaborators: Buffalo General Medical Center (Unknown); Erie County Medical Center (Other); Millard Fillmore Suburban Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: NB19-SSLHH-NA-FDA
Record Dates: First submitted 2021-07-28; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-07

CONDITIONS: Sepsis; Anemia; Bleeding; Erythrocytosis
Keywords: Lactate; Hemoglobin; Hematocrict
MeSH Terms: conditions — Sepsis; Anemia; Hemorrhage; Polycythemia | interventions — Hematocrit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Lactate, Hemoglobin, Hematocrit — Compare diagnostic tests to reference methods

SUMMARY:
The purpose of this study is to evaluate the clinical utility of the StatStrip Lactate, Hemoglobin and Hematocrit Hospital Meter System in the testing of whole blood specimens from patients in hospital settings by CLIA waived operators, over a period of at least twenty days. The specimens shall include capillary (obtained by fingerstick), and venous whole blood. The study will also evaluate the use of a Fingerstick Blood Contamination Barrier for capillary sampling from the fingertip. This submission to the FDA is intended for a Point of Care (POC), CLIA waived device for whole blood capillary and venous lactate, and hemoglobin and hematocrit measurements.

DETAILED DESCRIPTION:
The study will be conducted at three (3) different healthcare settings (hereafter referred to as "testing sites") in POC sites/departments, by at least nine (9) CLIAW operators (at least 3 in each healthcare setting), over a period of at least twenty days at each healthcare setting. Examples of hospital departments include (but are not limited to) Emergency Department (ED), Intensive Care Unit (ICU), Pediatric Intensive Care Unit (PICU), Surgical Intensive Care Unit (SICU), Medical Intensive Care Unit (MICU), Cardiac Intensive Care Unit (CICU), Operating Room (OR), where point-of-care lactate, hemoglobin and hematocrit testing can be utilized.

Each site will recruit at least 120 patients for a total of 360 adult patients in all three (3) sites for each of the tests and specimen types. An attempt will be made to enroll 50% males and 50% females.

Each Study Subject will provide:

1. Two (2) capillary whole blood fingerstick specimens

   1. One Lactate capillary test using the Fingerstick Blood Contamination Barrier
   2. One Hb/Hct capillary test following traditional fingerstick protocol
2. One (1) venous whole blood specimen obtained by venipuncture collected in a lithium heparin tube or heparinized syringe:

   1. One lactate venous test
   2. One Hb/Hct venous test

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (over or equal to 18 years old) with ordered hemoglobin and hematocrit

Exclusion Criteria:

* Pediatric

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Each site will recruit at least 120 patients for a total of 360 adult patients in all three (3) sites for each of the tests and specimen types. An attempt will be made to enroll 50% males and 50% females.
  Each Study Subject will provide:
  1. Two (2) capillary whole blood fingerstick specimens
     1. One Lactate capillary test using the Fingerstick Blood Contamination Barrier
     2. One Hb/Hct capillary test following traditional fingerstick protocol
  2. One (1) venous whole blood specimen obtained by venipuncture collected in a lithium heparin tube or heparinized syringe:
     1. One lactate venous test
     2. One Hb/Hct venous test
Sampling Method: Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Analytical verification of StatStrip Lactate, Hemoglobin and Hematocrit Hospital Meter System - Lactate comparison | 20 days
  StatStrip Lactate, Hemoglobin and Hematocrit Hospital Meter System, a point of care testing instrument is as effective as a reference laboratory method for Lactate blood results in mmol/L
Analytical verification of StatStrip Lactate, Hemoglobin and Hematocrit Hospital Meter System - Hemoglobin comparison | 20 days
  StatStrip Lactate, Hemoglobin and Hematocrit Hospital Meter System, a point of care testing instrument is as effective as a reference laboratory method for Hemoglobin blood results in g/dL
Analytical verification of StatStrip Lactate, Hemoglobin and Hematocrit Hospital Meter System - Hematocrit comparison | 20 days
  StatStrip Lactate, Hemoglobin and Hematocrit Hospital Meter System, a point of care testing instrument is as effective as a reference laboratory method for Hematocrit blood results in %

CONTACTS AND LOCATIONS:
Overall Officials: Brooke Lerner, PhD, FAEMS, Principal Investigator — Buffalo General Medical Center; Brooke Lerner, PhD, FAEMS, Principal Investigator — Erie County Medical Center; Brooke Lerner, PhD, FAEMS, Principal Investigator — Millard Fillmore Suburban Hospital
Locations (3):
- United States (3):
  - Buffalo General Medical Center, Buffalo, New York
  - Erie County Medical Center, Buffalo, New York
  - Millard Fillmore Suburban Hospital, Williamsville, New York

IPD SHARING:
Plan to Share IPD: No